CLINICAL TRIAL: NCT06172504
Title: Effect of Male Ejaculation Frequency on Semen Parameters
Brief Title: Ejaculation Frequency and Semen Parameters
Acronym: EFASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-HS-134
Record Dates: First submitted 2023-11-21; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Sperm; Fertility
Keywords: Semen Parameters; Ejaculation Frequency; the penultimate abstinence period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine whether the frequency of ejaculation in men had an effect on semen parameters.. The main questions it aims to answer are:

* question 1：Whether the frequency of ejaculation has an effect on semen parameters
* question 2：Whether the penultimate abstinence period has an effect on semen parameters

The participants were men who underwent semen examination in the andrology clinic of the Reproductive Center of the First Hospital of Jilin University. A brief medical history was collected from each volunteer, including demographic information, fertility history and as well as information regarding their general health.The focus of the investigation is the time of abstinence for this examination, the penultimate abstinence period, and the number of ejaculation since the last 1 month.

DETAILED DESCRIPTION:
The main subjects of this study were husbands who underwent semen examination, Including pre-conception, infertility, and his wife with a history of pregnancy loss. Before the examination, the basic information such as age, height, weight, smoking, drinking, infertility years, fertility and pregnancy history, marriage years, education, occupation and exclusion criteria have adverse effects on sperm were investigated.The focus of the investigation is the time of abstinence for this examination, the penultimate abstinence period, and the number of ejaculation since the last 1 month. According to World Health Organization standards, semen analysis requires abstinence for 48h to 7 days. Semen parameters were recorded, including sperm DNA fragmentation rate, sperm motility rate, total sperm count, sperm motility, and sperm morphology. The frequency of ejaculation was divided into four groups:(1)0-4 times/month;(2)5-8 times/month;(3) 8-12 times/month;(4) >12 times/month.

ELIGIBILITY:
Inclusion Criteria:

1. Normal ejaculation function, normal sexual life, masturbation can ejaculate
2. Male age between 22 and 45 years old.
3. According to World Health Organization standards, the semen examination time is within 48h to 7 days of abstinence.

Exclusion Criteria:

1. The man was diagnosed with extremely severe oligospermia (sperm concentration <1 million/ml) and azoospermia.
2. Identify the factors affecting semen parameters, long-term exposure to high temperature, long-term exposure to chemicals, heavy metals, radiation and other toxic and harmful substances, orchitis/epididymitis, cryptorchidism, radiotherapy and chemotherapy treatment, and taking drugs to improve sperm within three months

Ages: 22 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: The participants were men who underwent semen examination in the andrology clinic of the Reproductive Center of the First Hospital of Jilin University. Including pre-conception, infertility, and his wife with a history of pregnancy loss.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Effect of ejaculation frequency on sperm DNA fragmentation rate | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of sperm DNA fragment rate. Survey the basic information of the subjects and their frequency of ejaculation in the past month.The frequency of ejaculation was divided into four groups:(1) 0-4 times/month; (2) 5-8 times/month; (3) 8-12 times/month; (4) >12 times/month. The outcome was to compare whether there were differences in semen parameters between the groups
Effect of ejaculation frequency on sperm motility rate | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of sperm motility rate. Survey the basic information of the subjects and their frequency of ejaculation in the past month. The frequency of ejaculation was divided into four groups:(1) 0-4 times/month; (2) 5-8 times/month; (3) 8-12 times/month; (4) >12 times/month. The outcome was to compare whether there were differences in semen parameters between the groups
Effect of ejaculation frequency on total sperm count | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of total sperm count. Survey the basic information of the subjects and their frequency of ejaculation in the past month. The frequency of ejaculation was divided into four groups:(1) 0-4 times/month; (2) 5-8 times/month; (3) 8-12 times/month; (4) >12 times/month. The outcome was to compare whether there were differences in semen parameters between the groups
Effect of ejaculation frequency on sperm vitality rate | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of sperm vitality rate. Survey the basic information of the subjects and their frequency of ejaculation in the past month. The frequency of ejaculation was divided into four groups:(1) 0-4 times/month; (2) 5-8 times/month; (3) 8-12 times/month; (4) >12 times/month. The outcome was to compare whether there were differences in semen parameters between the groups
Effect of ejaculation frequency on sperm morphology | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of sperm morphology. Survey the basic information of the subjects and their frequency of ejaculation in the past month. The frequency of ejaculation was divided into four groups:(1) 0-4 times/month; (2) 5-8 times/month; (3) 8-12 times/month; (4) >12 times/month. The outcome was to compare whether there were differences in semen parameters between the groups

SECONDARY OUTCOMES:
Effect of the penultimate abstinence period on DNA fragmentation rate | 6 months
  The subjects abstained for 3-7 days and masturbated to collect semen for measurement of sperm morphology. Survey the basic information of the subjects and their penultimate abstinence period. The outcome was to compare whether the penultimate abstinence period had an effect on DNA fragmentation rate（the cutoff value is 15%). We plans to recruit more than 1000 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: yang yu, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Background] Vander Borght M, Wyns C. Fertility and infertility: Definition and epidemiology. Clin Biochem. 2018 Dec;62:2-10. doi: 10.1016/j.clinbiochem.2018.03.012. Epub 2018 Mar 16. PMID 29555319
- [Background] Leisegang K, Dutta S. Do lifestyle practices impede male fertility? Andrologia. 2021 Feb;53(1):e13595. doi: 10.1111/and.13595. Epub 2020 Apr 24. PMID 32330362
- [Background] Hanson BM, Aston KI, Jenkins TG, Carrell DT, Hotaling JM. The impact of ejaculatory abstinence on semen analysis parameters: a systematic review. J Assist Reprod Genet. 2018 Feb;35(2):213-220. doi: 10.1007/s10815-017-1086-0. Epub 2017 Nov 16. PMID 29143943
- [Background] Barbagallo F, Cannarella R, Crafa A, Manna C, La Vignera S, Condorelli RA, Calogero AE. The Impact of a Very Short Abstinence Period on Conventional Sperm Parameters and Sperm DNA Fragmentation: A Systematic Review and Meta-Analysis. J Clin Med. 2022 Dec 8;11(24):7303. doi: 10.3390/jcm11247303. PMID 36555920
- [Background] Stanford JB, White GL, Hatasaka H. Timing intercourse to achieve pregnancy: current evidence. Obstet Gynecol. 2002 Dec;100(6):1333-41. doi: 10.1016/s0029-7844(02)02382-7. PMID 12468181